CLINICAL TRIAL: NCT00358813
Title: An Open-Label, Non-Randomized, Pharmacokinetic and Safety Study of Multiple Oral Doses of GW679769 in Subjects With Renal Impairment
Brief Title: Observational Pharmacokinetic Study Of GW679769 In Subjects With Renal Impairment
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NKT102783
Record Dates: First submitted 2006-07-28; First posted 2006-08-01 (Estimated); Last update posted 2017-08-04 (Actual); Status verified 2017-08

CONDITIONS: Vomiting
Keywords: emesis; renal impairment; GW679769; kidney problems
MeSH Terms: conditions — Vomiting; Renal Insufficiency | interventions — casopitant

ARMS (1):
- Subjects receiving casopitant (Experimental): Eligible subjects will receive a 100 milligrams oral dose of casopitant once daily for five consecutive days.
  Interventions: Drug: Casopitant

INTERVENTIONS:
Drug: Casopitant — Casopitant oral tablets will be available with a dose of 50 milligrams.
  Other Names: GW679769

SUMMARY:
The purpose of the study is to evaluate how subjects with mild or moderate kidney problems process or breakdown the study drug GW679769 in their bodies as compared to healthy subjects.

ELIGIBILITY:
Inclusion criteria:

* Healthy or have mild or moderate renal impairment.
* Females must be of non-childbearing potential(hysterectomy, bilateral oophorectomy, post-menopausal) OR childbearing and must have a negative pregnancy test and meet/comply with one of the following: abstinence, double-barrier contraception, vasectomized partner).
* Be negative for Hepatitis B and C.
* Have negative results on drug, alcohol and HIV tests.
* Have stable renal function.

Exclusion criteria:

* Have a peptic ulcer.
* Abuse drugs or alcohol.
* Are pregnant or lactating.
* Have heart failure.
* Have uncontrolled emesis.
* Have an infection.
* Have taken or received inducers or inhibitors of CYP3A4 or CYP3A5 within 14 days of study start.
* Active peptic ulcer disease.
* Digoxin use.
* Laboratory results that show low iron or pepsinogen levels, AST and CK level >1,5 ULN, or that show stool is positive for occult blood.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2006-09-08 (Actual); Primary Completion 2008-08-22 (Actual); Study Completion 2008-08-22 (Actual)

PRIMARY OUTCOMES:
Area under the plasma drug concentration versus time curve from 0 to 24 hours (AUC[0-24]) of casopitant and GSK525060 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 16 hours on Day 1; pre-dose on Day 2, Day 3 and Day 4; Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours on Day 5
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Maximum observed concentration (Cmax) of casopitant and GSK525060 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 16 hours on Day 1; pre-dose on Day 2, Day 3 and Day 4; Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours on Day 5
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.

SECONDARY OUTCOMES:
Time to maximum observed plasma drug concentration (Tmax) of casopitant and GSK525060 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 16 hours on Day 1; pre-dose on Day 2, Day 3 and Day 4; Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours on Day 5
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Half-life of casopitant and GSK525060 | Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12 and 16 hours on Day 1; pre-dose on Day 2, Day 3 and Day 4; Pre-dose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 6, 8, 10, 12, 16, 24, 36, and 48 hours on Day 5
  Blood samples will be collected at the indicated time points for pharmacokinetic analysis.
Free fraction (percent unbound) of casopitant and GSK525060 | 1,2,4 and 24 hours post-dose on Day 1; pre-dose,1,2,4 and 24 hours post-dose on Day 5
  Blood samples will be collected for assessment of protein binding of casopitant and GSK525060.
Number of subjects with adverse events (AEs) and serious adverse events (SAEs) | Up to Day 22
  An AE is any untoward medical occurrence in a subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. Any untoward event resulting in death, life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, congenital anomaly/birth defect or any other situation according to medical or scientific judgment will be categorized as SAE.
Number of subjects with abnormal values for blood pressure | Up to Day 22
  Systolic (SBP) and diastolic blood pressure (DBP) will be measured.
Number of subjects with abnormal values for heart rate | Up to Day 22
  Heart rate will be measured.
Number of subjects with abnormal findings after weight measurement | Up to Day 22
  Weight evaluation will be performed as measure of safety.
Number of subjects having abnormal hematology laboratory parameters as a measure of safety | Up to Day 22
  Hematology parameters will be analyzed as a measure of safety.
Number of subjects having abnormal clinical Chemistry laboratory parameters as a measure of safety | Up to Day 22
  Clinical chemistry parameters will be analyzed as a measure of safety.
Number of subjects having abnormal values for urinalysis as a measure of safety | Up to Day 22
  Urinalysis will be carried out as a measure of safety.
Number of subjects with abnormal findings after serological tests | Up to Day 22
  Serological tests will be performed as a measure of safety.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (3):
- United States (3):
  - GSK Investigational Site, Miramar, Florida
  - GSK Investigational Site, Orlando, Florida
  - GSK Investigational Site, Minneapolis, Minnesota

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- See also: Results for study NKT102783 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/NKT102783?search=study&study_ids=NKT102783#rs
- Available data/document: Annotated Case Report Form: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKT102783 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register